CLINICAL TRIAL: NCT02440828
Title: Ventilator Associated Pneumonia: Addition of Tobramycin Inhalation Antibiotic Treatment to Standard IV Antibiotic Treatment
Brief Title: Addition of Tobramycin Inhalation in the Treatment of Ventilator Associated Pneumonia
Acronym: VAPORISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, R.A.S. Hoek, MD, MD, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VAP-2014; 2014-001406-17 (EudraCT Number)
Record Dates: First submitted 2015-03-13; First posted 2015-05-12 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Ventilator Associated Pneumonia (VAP)
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tobramycin inhalation (Experimental): twice daily tobramycin inhalation (Bramitob) 300 mg and standard intravenous antibiotics treatment
  Interventions: Drug: tobramycin inhalation
- Placebo (Placebo Comparator): twice daily placebo inhalation and standard intravenous antibiotics treatment
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tobramycin inhalation — tobramycin inhalation 300 mg twice daily
  Other Names: Bramitob
  Arms: tobramycin inhalation
Drug: placebo — NaCl 0.9% inhalation 4 ml twice daily
  Other Names: NaCl 0.9% inhalation 4 ml
  Arms: Placebo

SUMMARY:
This study evaluates the addition of tobramycin inhalation treatment to standard intravenous therapy in the treatment of ventilator associated pneumonia.

DETAILED DESCRIPTION:
Rationale: Approximately 9-27% of mechanically ventilated patients in the intensive care unit (ICU) develop ventilator-associated pneumonia (VAP). Patients in whom VAP develops have a higher mortality rate up to 50%, stay longer in the intensive care unit (ICU), and require more resources than those without the disease. Despite the availability of modern ICU care and modern antibiotics, the overall clinical cure rate after 72 hours of antibiotic treatment for VAP is only 40%. The cure rate for Pseudomonas aeruginosa is even lower. It is unclear why VAP cure rates are so low. The ATS guidelines recommend IV antibiotic treatment (IV AB), especially directed against gram-negative microorganisms. However, the relatively poor response rates seen with intravenous therapy of VAP and the emergence of MDR organisms makes new treatment options desirable. The ATS/IDSA VAP guidelines recommend that "adjunctive therapy with an inhaled aminoglycoside or polymyxin (colistin) for MDR Gram-negative pneumonia should be considered, especially in patients who are not improving". It is therefore necessary to investigate whether adjunctive therapy with inhalation Tobramycin could ameliorate prognosis. The recommendations by the Society of Infectious Diseases Pharmacists are similar.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation 48 hours or more
* New or progressive radiologic pulmonary infiltrate

Together with at least two of the following three criteria (< 24 h):

* temperature >38°C
* leukocytosis >12,000/mm3 or leucopenia <4,000/mm3
* purulent respiratory secretions

Exclusion Criteria:

* patients with allergy to tobramycin
* pregnancy
* expected to die within 72 hours after enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-03; Primary Completion 2020-03-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
response after 72 h of treatment | 72 hours
  non response is considered when at least one of the following is present
  1. No improvement of the arterial O2 tension to inspired O2 fraction ratio
  2. Persistence of fever (≥38°C) or hypothermia (<35.5°C) together with purulent respiratory secretions
  3. increase in the pulmonary infiltrates on chest radiograph of greater than or equal to 50%
  4. occurrence of septic shock or multiple organ dysfunction syndrome, defined as three or more organ system failures not present on Day 1

SECONDARY OUTCOMES:
Mortality rate | day 30
  30-day and 90- day mortality rate
Mortality rate | day 90
  30-day and 90- day mortality rate
ICU survival | day 90
Absence of hospital admittance at day 60 | day 60
Discharge from the ICU | up to 60 days
  Patients will be followed during ICU stay and evaluated at discharge from ICU, expected average time of discharge is 10 days
Ventilator free days at day 28 | up to 28 days
Adverse events | day 1
Adverse events | day 4
Adverse events | day 8
Adverse events | day 14
Adverse events | day 30
Adverse events | day 90
Day of normalisation of CRP | day 1
Day of normalisation of CRP | day 4
Day of normalisation of CRP | day 8
Day of normalisation of CRP | day 14
Day of normalisation of CRP | day 30
Day of normalisation of CRP | day 90
Eradication of pathogens | day 4
Eradication of pathogens | day 8
Eradication of pathogens | day 14
Eradication of pathogens | day 30
Eradication of pathogens | day 90
Clinical Pulmonary Infectious Score (CPIS) | Day 1
Clinical Pulmonary Infectious Score (CPIS) | Day 4
Clinical Pulmonary Infectious Score (CPIS) | Day 8
Clinical Pulmonary Infectious Score (CPIS) | Day 14
Clinical Pulmonary Infectious Score (CPIS) | discharge ICU, expected average time of discharge is 10 days
APACHE II score | Day 1
APACHE II score | Day 4
APACHE II score | Day 8
APACHE II score | Day 14
APACHE II score | discharge ICU, expected average time of discharge is 10 days
Multiple Organ Dysfunction score (MODS) | Day 1
Multiple Organ Dysfunction score (MODS) | Day 4
Multiple Organ Dysfunction score (MODS) | Day 8
Multiple Organ Dysfunction score (MODS) | Day 14
Multiple Organ Dysfunction score (MODS) | discharge ICU, expected average time of discharge is 10 days
Sequential Organ Failure Assessment score (SOFA) | Day 1
Sequential Organ Failure Assessment score (SOFA) | Day 4
Sequential Organ Failure Assessment score (SOFA) | Day 8
Sequential Organ Failure Assessment score (SOFA) | Day 14
Sequential Organ Failure Assessment score (SOFA) | discharge ICU, expected average time of discharge is 10 days
Lung Injury Score (LIS) | Day 1
Lung Injury Score (LIS) | Day 4
Lung Injury Score (LIS) | Day 8
Lung Injury Score (LIS) | Day 14
Lung Injury Score (LIS) | discharge ICU, expected average time of discharge is 10 days
Day of normalisation of procalcitonin (PCT) | day 1
Day of normalisation of procalcitonin (PCT) | day 4
Day of normalisation of procalcitonin (PCT) | day 8
Day of normalisation of procalcitonin (PCT) | day 14
Day of normalisation of procalcitonin (PCT) | day 30
Day of normalisation of procalcitonin (PCT) | day 90
Day of normalisation of chest X-ray | day 1
Day of normalisation of chest X-ray | day 4
Day of normalisation of chest X-ray | day 8
Day of normalisation of chest X-ray | day 14
Day of normalisation of chest X-ray | day 30
Day of normalisation of chest X-ray | day 90

CONTACTS AND LOCATIONS:
Overall Officials: Menno Van der Eerden, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (2):
- Erasmus MC, Rotterdam, Netherlands
- Hospital Clinic, Barcelona, Spain